CLINICAL TRIAL: NCT01867281
Title: The Effect of Aspirin Desensitization on Patients With Aspirin-exacerbated Respiratory Diseases
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: Rassoul Akram Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 92-01-119-20728
Record Dates: First submitted 2013-05-29; First posted 2013-06-03 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Asthma, Aspirin-Induced
Keywords: aspirin; asthma; Aspirin desensitization; Aspirin induced asthma; Immune System Diseases; Respiratory Hypersensitivity
MeSH Terms: conditions — Asthma, Aspirin-Induced; Asthma; Immune System Diseases; Respiratory Hypersensitivity | interventions — Aspirin

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention: Aspirin (Active Comparator): Participants will undergo aspirin desensitization over a 2-day period with increasing doses of aspirin (60, 125, 325 and 625 mg). Thereafter,they will be followed with 625 mg aspirin bid.
  Interventions: Drug: aspirin
- Control: placebo (Placebo Comparator): Participants will receive placebo

INTERVENTIONS:
Drug: aspirin
  Arms: Intervention: Aspirin

SUMMARY:
The purpose of this study is to determine the effect of aspirin desensitization on symptoms and immunologic profile of patients with aspirin-exacerbated respiratory diseases (AERD).

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical diagnose of aspirin-exacerbated respiratory disease
* History of physician diagnosed asthma.
* History of physiacian diagnosed chronic rhinosinositis with nasal polyps.
* Positive reaction to aspirin challenge test.
* Stable asthma (post-bronchodilator FEV1 of 70% or better, no increase in baseline dose of oral glucocorticoids for at least 3 months, and no history of hospitalization or emergency room visits for asthma for at least the prior 6 months).

Exclusion Criteria:

* Being smoker
* pregnancy
* Current breastfeeding
* History of bleeding diathesis
* History of transient ischemic attack or stroke, or diabetes.
* History of abnormal hepatic function
* Uncontrolled hypertension or use of beta blocker medication.
* History of gastrointestinal ulcers or gastrointestinal bleeding.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in SNOT-22 scores from Baseline | 6 months
  At baseline and 6 months after treatment, all participants will complete the SNOT-22 questionnaire. SNOT-22 is a validated disease specific questionnaire that assesses the health related quality of life patients.
change in serum concentration of IL-10 | 6 months
  At baseline and 6 months after treatment, serum level of IL-10 will be investigated for all participants.
change in concentration of serum TGF-beta | 6 months
  At baseline and 6 months after treatment, serum level of TGF-beta will be investigated for all participants
change in concentration of serum IFN-gamma | 6 months
  At baseline and 6 months after treatment, serum level of IFN-gamma will be investigated for all participants.

SECONDARY OUTCOMES:
Lund Mackay score | 6 months
  For all participants, Lund Mackay will be scored by investigators.
Asthma attacks | 6 months
  Number of asthma attacks will be recorded for all participants over a 6-month follow up.
medication needs | 6 months
  Medication needs to relief respiratory symptoms will be recorded for all participants over a 6-month period.
FEV1 | 6 months
  FEV1 for all patients will be assessed using spirometery

CONTACTS AND LOCATIONS:
Overall Officials: Hossein Esmaeilzadeh, MD, Study Director — Department of Allergy and Immunology, Rasool-e-Akram Hospital, Tehran University of Medical Sciences.; Mohammad Nabavi, MD, Study Chair — Department of Allergy and Immunology, Rasool-e-Akram Hospital, Tehran University of Medical Sciences.; Zahra Aryan, MD, MPH, student, Principal Investigator — Molecular Immunology Research Center, Tehran University of Medical Sciences.
Locations (1):
- Department of Allergy and Immunology, Rasool-e-Akram Hospital, Tehran University of Medical Sciences, Tehran, Tehran Province, Iran

REFERENCES:
- [Background] Katial RK, Strand M, Prasertsuntarasai T, Leung R, Zheng W, Alam R. The effect of aspirin desensitization on novel biomarkers in aspirin-exacerbated respiratory diseases. J Allergy Clin Immunol. 2010 Oct;126(4):738-44. doi: 10.1016/j.jaci.2010.06.036. Epub 2010 Aug 21. PMID 20728206
- [Background] White AA, Stevenson DD. Does suppression of IL-4 synthesis by aspirin explain the therapeutic benefit of aspirin desensitization treatment? J Allergy Clin Immunol. 2010 Oct;126(4):745-6. doi: 10.1016/j.jaci.2010.08.037. No abstract available. PMID 20920763
- [Background] Rozsasi A, Polzehl D, Deutschle T, Smith E, Wiesmiller K, Riechelmann H, Keck T. Long-term treatment with aspirin desensitization: a prospective clinical trial comparing 100 and 300 mg aspirin daily. Allergy. 2008 Sep;63(9):1228-34. doi: 10.1111/j.1398-9995.2008.01658.x. PMID 18699939
- [Background] Menzies D, Nair A, Meldrum KT, Hopkinson P, Lipworth BJ. Effect of aspirin on airway inflammation and pulmonary function in patients with persistent asthma. J Allergy Clin Immunol. 2008 May;121(5):1184-1189.e4. doi: 10.1016/j.jaci.2008.01.009. Epub 2008 Mar 4. PMID 18313127
- [Background] Swierczynska M, Nizankowska-Mogilnicka E, Zarychta J, Gielicz A, Szczeklik A. Nasal versus bronchial and nasal response to oral aspirin challenge: Clinical and biochemical differences between patients with aspirin-induced asthma/rhinitis. J Allergy Clin Immunol. 2003 Nov;112(5):995-1001. doi: 10.1016/s0091-6749(03)02015-3. PMID 14610494
- [Background] Vaidyanathan S, Williamson PA, Lipworth BJ. Is a positive nasal lysine-aspirin challenge test associated with a more severe phenotype of chronic rhinosinusitis and asthma? Am J Rhinol Allergy. 2012 May-Jun;26(3):e89-93. doi: 10.2500/ajra.2012.26.3767. PMID 22643934
- [Background] Higashi N, Taniguchi M, Mita H, Yamaguchi H, Ono E, Akiyama K. Aspirin-intolerant asthma (AIA) assessment using the urinary biomarkers, leukotriene E4 (LTE4) and prostaglandin D2 (PGD2) metabolites. Allergol Int. 2012 Sep;61(3):393-403. doi: 10.2332/allergolint.11-RA-0403. Epub 2012 May 25. PMID 22627848
- [Background] Chang JE, White A, Simon RA, Stevenson DD. Aspirin-exacerbated respiratory disease: burden of disease. Allergy Asthma Proc. 2012 Mar-Apr;33(2):117-21. doi: 10.2500/aap.2012.33.3541. PMID 22525387